CLINICAL TRIAL: NCT04091581
Title: Comparison of Tear Evaporation Rate With Systane Complete in Dry Eye and Non-Dry Eye
Acronym: BULLDOG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 41327
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Results first posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Evaporative Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Non-Dry Eye (Experimental): Instill eye drop and perform followup assessments on people with a Ocular Surface Disease Index score <13 and a non-invasive Keratograph break-up time of >/= 10 seconds in the worst eye
  Interventions: Drug: Systane Complete
- Dry Eye (Experimental): Instill eye drop and perform followup assessments on people with an Ocular Surface Disease Index score >/= 13 and a non-invasive Keratograph break-up time </= 5 seconds in the worst eye
  Interventions: Drug: Systane Complete

INTERVENTIONS:
Drug: Systane Complete — Systane Complete will be instilled and rate of evaporation assessed before and after.

SUMMARY:
The objective of the study is to compare the rate of tear evaporation, measured with a novel evaporimeter, before and for one hour after an eye drop containing nano-sized oil droplets has been instilled.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Is willing to be awake for at least 2 hours before visit 2;
5. Is willing not to wear eye makeup on the day of visit 2;
6. Is willing not to use eye drops or artificial tears on the days of visits 1 or 2;
7. Group specific criteria:

   1. Dry eye participant group: Symptoms: OSDI ≥ 13 and Signs: NIKBUT ≤ 5 s in the worst eye
   2. Non-dry eye participant group: Symptoms: OSDI < 13 and Signs: NIKBUT ≥ 10 s in the worst eye

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to sodium fluorescein dye;
6. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit);
7. Is aphakic;
8. Has undergone refractive error surgery;
9. Has undergone ocular surgery in the last 6 months;
10. Has punctal plugs;
11. Has a known sensitivity to Systane eye drops (including Systane Balance, Systane Complete, Systane Gel Drops, Systane Ultra, etc.)
12. Has a known sensitivity to petroleum jelly (Vaseline);
13. Has epilepsy and/or sensitivity to flashing lights;
14. Has worn contact lenses within the past month or is planning to wear contact lenses during the study;
15. Has any physical impairment that would interfere with holding the evaporimeter;
16. Has taken part in another clinical research study involving ocular drops or treatments within the last 14 days; * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — Centre for Ocular Research & Education
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a single study center located in Canada.
Groups:
- Non-Dry Eye: Tear evaporation was measured prior to and after a single 15 µl instillation of Systane Complete was instilled in people with an Ocular Surface Disease Index score <13 and a non-invasive Keratograph break-up time >/= 10 seconds in the worst eye.
- Dry Eye: Tear evaporation was measured prior to and after a single 15 µl instillation of Systane Complete in people with an Ocular Surface Disease Index score >/= 13 and a non-invasive Keratograph break-up time </= 5 seconds in the worst eye.
Period: Overall Study
Arm/Group | Non-Dry Eye | Dry Eye
Started | 10 | 11
Completed | 10 | 10
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Non-Dry Eye; Dry Eye: Tear evaporation was measured prior to and after Systane Complete was instilled.
- Total: Total of all reporting groups
Arm/Group | Non-Dry Eye | Dry Eye | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (12.8) | 45.4 (22.7) | 39.3 (19.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 3 | 1 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Tear Evaporation Rate
Description: Tear film evaporation rate (% relative humidity per second) was performed using a novel evaporimeter as a non-invasive measurement of tear film evaporation. The slope was calculated from the change in humidity between 7 to 17.5 seconds while the eye was open and between 10 to 17.5 seconds when the eye was closed. Data from the right eye was analyzed.
Time Frame: Baseline (Prior to instillation); 10, 30 and 60 minutes post instillation of eye drop
Population: The analysis population includes all participants that were exposed to Systane Complete, and excludes the one dry eye subject that was lost to follow-up.
Measure: Mean (Standard Deviation); unit: % relative humidity per second
Groups:
- Non-Dry Eye: Tear evaporation was measured prior to and after Systane Complete was instilled in people without dry eye.
- Dry Eye: Tear evaporation was measured prior to and after Systane Complete was instilled in people with dry eye.
Arm/Group | Non-Dry Eye | Dry Eye
Number analyzed (Participants) | 10 | 10
% relative humidity per second
  Baseline | 1.15 (0.19) | 1.38 (0.22)
  10 minutes post-drop | 1.26 (0.31) | 1.32 (0.25)
  30 minutes post-drop | 1.01 (0.24) | 1.18 (0.27)
  60 minutes post-drop | 1.07 (0.31) | 1.27 (0.27)
Statistical Analysis 1: Comparison: Non-Dry Eye; Test type: Other; p = 0.002, ANOVA
Statistical Analysis 2: Comparison: Non-Dry Eye vs Dry Eye; Comparison of the baseline tear evaporation rate of the non-dry eye and dry eye group; Test type: Other; p = 0.022, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent for the duration of the study (up to 2 weeks). Adverse events are reported as pre-treatment or post-treatment.
Description: An adverse event was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, whether or not related to the medical device.
Groups:
- Non-Dry Eye: Tear evaporation was measured prior to and after Systane Complete was instilled in a group of people without dry eye that had an Ocular Surface Disease Index score <13 and a non-invasive Keratograph break-up time >/= 10 seconds in the worst eye.
- Dry Eye: Tear evaporation was measured prior to and after Systane Complete was instilled in a group of people with dry eye that had an Ocular Surface Disease Index score >/=13 and a non-invasive Keratograph break-up time </= 5 seconds in the worst eye.
Arm/Group | Non-Dry Eye | Dry Eye
All-Cause Mortality (participants affected / at risk) | 1/10 | 2/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 1/10 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Dry Eye (N=10) | Dry Eye (N=11)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Steroid injection (Surgical and medical procedures) | 0 (0) | 1 (1)
Common cold (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT04091581/Prot_SAP_000.pdf